CLINICAL TRIAL: NCT02548936
Title: Efficacy and Safety of Simvastatin-ezetimibe Combination Therapy in Reduction of Progression of Atherosclerosis Among Patients With Systemic Lupus Erythematosus: A Randomized Single-Blind Trial
Brief Title: Efficacy and Safety of Simvastatin-ezetimibe Combination Therapy Among Patients With SLE
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: pumch-sleas
Record Dates: First submitted 2015-08-31; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-08

CONDITIONS: Atherosclerosis
Keywords: Cholesterol, LDL; Carotid Intima-Media Thickness; Atherosclerosis; Ezetimibe, Simvastatin Drug Combination; Lupus Erythematosus, Systemic
MeSH Terms: conditions — Atherosclerosis; Lupus Erythematosus, Systemic | interventions — Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipid-lowering treatment (Experimental): The Lipid-lowering treatment is Ezetimibe+Simvastatin Drug Combination by oral administration. The patients in intervention group received simvastatin (10mg/day) + ezetimibe (20 mg/day) combined therapy for 12 month.
  Interventions: Drug: Ezetimibe+Simvastatin Drug Combination
- No lipid-lowering treatment (No Intervention): Without any Lipid-lowering treatment for 12 month.

INTERVENTIONS:
Drug: Ezetimibe+Simvastatin Drug Combination — The patients in Ezetimibe+Simvastatin Drug Combination group received simvastatin (10mg/day) + ezetimibe (20 mg/day) by oral administration for 12 month.
  Other Names: ezetimibe/simvastatin
  Arms: Lipid-lowering treatment

SUMMARY:
This is a randomized single-blind trial. This study aimed to determine if intensive lipid-lowering therapy (simvastatin-ezetimibe combination therapy) could reduce the progression of atherosclerosis effectively and safely among SLE patients with carotid artery intima thickening. The study results were expected to be helpful for SLE patients in preventing atherosclerosis.

DETAILED DESCRIPTION:
Patient Registries: A convenient consecutive sampling was used to recruit participants from outpatients in department of rheumatism of PUMCH. Prior to their enrollment in the study, all patients gave written, informed consent. To minimize subject non-response or rejection, the investigators inform patients the benefits and risks, and feedback them all physical examination results for free in the recruit period.

Randomization: A randomization will be used to allocate patients into Lipid-lowering treatment group and control group.

Blind: A trained ultrasonographer who assessed carotid intima media thickness (CIMT) (at baseline and 12 months) will be blinded to all clinical and treatment information.

Statistical analysis: The characteristics of the study sample were summarized using descriptive statistics with dichotomous or ordinal data presented as percentages and continuous data as means, standard deviations, and medians, interquartile range. Differences of progression rate of atherosclerosis between intervention group and control group were assessed with either the t test or the non-parametric Wilcoxon test. A multivariable linear regression model will be used to evaluate the relationship between the progression of CIMT and intervention after controlling for confounding factors. Statistical significance was defined as a 2-tailed P value less than 0.05. All calculations were performed using SAS version 9.3.

Quality Control and Data Management: Two doctors (not the main investigator) who come from department of cardiology with the experiences of clinical trial and a data manager will be serving as Data and Safety Monitor. A monthly meeting will be set up for investigators and monitors. The monitors need to review the study protocol and set Data Safety Management plan before recruitment. Then, they need to review rates of recruitment, adherence, follow-up conditions and assess the efficacy and harm during the study. If Monitors find that the simvastatin-ezetimibe combination therapy is causing severe adverse event, then a detailed record is needed. Monitors need to inform the main investigator within 3 hours and to inform state China Food and Drug Administration within 24 hours. Interim monitoring will focus on data quality, percentage of AE or SAE, and evidence of benefit.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years and clinical diagnosis of SLE
2. abnormal CIMT (≥0.9 mm at any site) by B-mode ultrasound
3. LDL-C≥100mg/dl
4. a signed written informed consent was able to be obtained.

Exclusion Criteria:

1. atherosclerotic cardiovascular disease
2. diabetes
3. history of intolerance or allergy to the statins or ezetimibe
4. had ever received statins or ezetimibe within 12 months of study entry
5. LDL-C≥190mg/dl
6. active infection
7. ALT was higher than 2 times of the upper normal limit or CK was higher than 1.5 times of the upper normal limit.
8. pregnant or lactating women
9. patients with severe SLE.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The change of carotid intima media thickness over 12 months | baseline, 12 months
  CIMT(Unit: millimeter) is defined as the distance between the lumen-intima interface and the media-adventitia interface, which corresponded to the inner and outer echogenic lines seen on the B-mode ultrasound image.

SECONDARY OUTCOMES:
The rate of abnormal elevated alanine aminotransferase (ALT) | 1 month
  ALT >40U/L
The rate of abnormal elevated alanine aminotransferase | 3 months
  ALT >40U/L
The rate of abnormal elevated alanine aminotransferase | 6 months
  ALT >40U/L
The rate of abnormal elevated alanine aminotransferase | 12 months
  ALT >40U/L
The rate of abnormal elevated creatine kinase (CK) | 1 month
  CK >60U/L
The rate of abnormal elevated creatine kinase | 3 month
  CK >60U/L
The rate of abnormal elevated creatine kinase | 6 month
  CK >60U/L
The rate of abnormal elevated creatine kinase | 12 month
  CK >60U/L

CONTACTS AND LOCATIONS:
Overall Officials: Shuyang Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China